CLINICAL TRIAL: NCT01933581
Title: ICON1: A Study to Improve Cardiovascular Outcomes in High Risk PatieNts With Acute Coronary Syndrome
Brief Title: A Study to Improve Cardiovascular Outcomes in High Risk PatieNts With Acute Coronary Syndrome
Acronym: ICON1
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 12742
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACS undergoing CA and PCI: Patients with Acute Coronary Syndrome undergoing coronary angiography and PCI

SUMMARY:
Coronary artery disease and heart attacks are the leading cause of death in the UK. Our population is ageing. The number of older patients suffering heart attacks and having angioplasty procedures to open up blocked heart arteries is increasing. After angioplasty, older patients (80 years of age or over) are at 5 times increased risk of death at one year compared to their predicted normal life expectancy. In addition, many patients present with further heart attacks, stroke and undergo repeat heart catheter test and angioplasty procedures. At present it is not clear who will or will not experience further problems in the future. The ability to predict who will and will not suffer future problems at the time of initial presentation can be helpful in providing additional treatment and close monitoring to those that are at risk of further problems. The ICON 1 study is set out to study just that. In this study, older patients will undergo a comprehensive evaluation of the cardiovascular disease burden by undergoing additional investigations. These results from each patient will be used to develop a risk score that will inform physicians of the patient's future risk of developing adverse events and provide a better understanding of how to manage older patients with coronary artery disease and also help plan future studies looking at treatment strategies that might be beneficial in improving outcomes.

ELIGIBILITY:
Inclusion criteria: Older patients (65+) presenting with ACS for coronary angiography will be recruited into this study.

Exclusion criteria: Those presenting with cardiogenic shock, those with co-existing malignancy with life expectancy less than one year and those with evidence of active infection such as urinary tract infection, pneumonia, sepsis and any wound infection will also be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: ICON 1 is a prospective cohort study of older patients presenting with ACS.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Composite outcome: occurrence of one or more of death, myocardial infarction, stroke, repeat revascularisation, Bleeding Academic Research Consortium (BARC) defined bleeding | 1 YEAR

SECONDARY OUTCOMES:
Quality of life SF 36, EQ 5D | 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Kunadian, MD FRCP, Principal Investigator — Newcastle University and NUTH NHS Trust
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Rubino F, Brugaletta S, Mills G, Pompei G, Scarsini R, Ribichini F, Raber L, Kunadian V. Coronary Artery Plaque Phenotype and 5-Year Clinical Outcomes in Older Patients with Non-ST Elevation Acute Coronary Syndrome. Rev Cardiovasc Med. 2024 May 14;25(5):168. doi: 10.31083/j.rcm2505168. eCollection 2024 May. PMID 39076483
- [Derived] Dirjayanto VJ, Martin-Ruiz C, Pompei G, Rubino F, Kunadian V. The association of inflammatory biomarkers and long-term clinical outcomes in older adults with non-ST elevation acute coronary syndrome. Int J Cardiol. 2024 Aug 15;409:132177. doi: 10.1016/j.ijcard.2024.132177. Epub 2024 May 16. PMID 38761976
- [Derived] Dirjayanto VJ, Pompei G, Rubino F, Biscaglia S, Campo G, Mihailidou AS, den Ruijter H, Kunadian V. Non-invasive vascular measures as prognostic predictors for older patients with non-ST elevation acute coronary syndrome. Coron Artery Dis. 2024 Aug 1;35(5):368-381. doi: 10.1097/MCA.0000000000001352. Epub 2024 Mar 4. PMID 38436050
- [Derived] Dirjayanto VJ, Alkhalil M, Dodson J, Mills G, Pompei G, Rubino F, Kunadian V. Cognitive impairment and outcomes in older adults with non-ST-elevation acute coronary syndrome. Heart. 2024 Feb 23;110(6):416-424. doi: 10.1136/heartjnl-2023-323224. PMID 37813562
- [Derived] Ratcovich H, Beska B, Mills G, Holmvang L, Adams-Hall J, Stevenson H, Veerasamy M, Wilkinson C, Kunadian V. Five-year clinical outcomes in patients with frailty aged >/=75 years with non-ST elevation acute coronary syndrome undergoing invasive management. Eur Heart J Open. 2022 May 16;2(3):oeac035. doi: 10.1093/ehjopen/oeac035. eCollection 2022 May. PMID 35919345
- [Derived] Beska B, Mills GB, Ratcovich H, Wilkinson C, Damluji AA, Kunadian V. Impact of multimorbidity on long-term outcomes in older adults with non-ST elevation acute coronary syndrome in the North East of England: a multi-centre cohort study of patients undergoing invasive care. BMJ Open. 2022 Jul 26;12(7):e061830. doi: 10.1136/bmjopen-2022-061830. PMID 35882457
- [Derived] Beska B, Coakley D, MacGowan G, Adams-Hall J, Wilkinson C, Kunadian V. Frailty and quality of life after invasive management for non-ST elevation acute coronary syndrome. Heart. 2022 Feb;108(3):203-211. doi: 10.1136/heartjnl-2021-319064. Epub 2021 May 14. PMID 33990413
- [Derived] Chan D, Martin-Ruiz C, Saretzki G, Neely D, Qiu W, Kunadian V. The association of telomere length and telomerase activity with adverse outcomes in older patients with non-ST-elevation acute coronary syndrome. PLoS One. 2020 Jan 10;15(1):e0227616. doi: 10.1371/journal.pone.0227616. eCollection 2020. PMID 31923255
- [Derived] Gu SZ, Qiu W, Batty JA, Sinclair H, Veerasamy M, Brugaletta S, Neely D, Ford G, Calvert PA, Mintz GS, Kunadian V. Coronary artery lesion phenotype in frail older patients with non-ST-elevation acute coronary syndrome undergoing invasive care. EuroIntervention. 2019 Jun 12;15(3):e261-e268. doi: 10.4244/EIJ-D-18-00848. PMID 30777840
- [Derived] Gu SZ, Beska B, Chan D, Neely D, Batty JA, Adams-Hall J, Mossop H, Qiu W, Kunadian V. Cognitive Decline in Older Patients With Non- ST Elevation Acute Coronary Syndrome. J Am Heart Assoc. 2019 Feb 19;8(4):e011218. doi: 10.1161/JAHA.118.011218. PMID 30773118
- [Derived] Kunadian V, Neely RD, Sinclair H, Batty JA, Veerasamy M, Ford GA, Qiu W. Study to Improve Cardiovascular Outcomes in high-risk older patieNts (ICON1) with acute coronary syndrome: study design and protocol of a prospective observational study. BMJ Open. 2016 Aug 23;6(8):e012091. doi: 10.1136/bmjopen-2016-012091. PMID 27554105
- [Derived] Sinclair H, Batty JA, Qiu W, Kunadian V. Engaging older patients in cardiovascular research: observational analysis of the ICON-1 study. Open Heart. 2016 Aug 3;3(2):e000436. doi: 10.1136/openhrt-2016-000436. eCollection 2016. PMID 27547431